CLINICAL TRIAL: NCT07249970
Title: Trajectories of People With Substance or Behavioral Addictions in Contact With the Healthcare System: Medical, Neurobiological, Sociological, and Psychological Characteristics. Multicenter, Multidisciplinary Prospective Study.
Brief Title: Understanding the Long-term Paths of People With Addictions
Acronym: ADDICT AQUI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-20 ADDICTAQUI; CCPPRB BORDEAUX B (Other: Ethic Committee)
Record Dates: First submitted 2025-09-29; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Addiction Disorders; Addictive Behaviors; Addiction
Keywords: Addiction; addictive behavior; addiction disorders
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual care
  Interventions: Other: Addiction Severity Index

INTERVENTIONS:
Other: Addiction Severity Index — Once recruited, self-questionnaires completed by the participant at home and brought back at next visite, during which the participant takes cognitive tests. Follow-up interviews are scheduled at 3 months, 6 months, and then every 6 months.

SUMMARY:
The study is an open prospective cohort study. Participants are assessed at the start of their care in an addiction treatment unit using the Addiction Severity Index (ASI) and the Mini International Neuropsychiatric Interview (MINI), which are routinely conducted in these centers for individuals with substance use or behavioral disorders. After the study protocol is explained, the evaluator checks eligibility criteria, interested participants provide their written informed consent. The evaluator invites participants to complete self-administered questionnaires at home, which are returned during a session that also includes cognitive testing. Follow-up interviews are scheduled at 3 months, 6 months, and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for substance or behavioral addiction at one of the inclusion centers, with more than one month to wait before treatment begins
* Presenting with at least one substance or behavioral addiction (according to DSM5 criteria)

Exclusion Criteria:

* Condition incompatible with understanding assessment tools
* Difficulties understanding and/or writing French
* Person unable to give personal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare units : CSAPA de Bordeaux and CSAPA de Bayonne.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2002-03-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of addiction | at Day 0, at Month 3, at Month 6 and at each following 6-month visit
  ASI composite score

CONTACTS AND LOCATIONS:
Overall Officials: Marc AURIACOMBE, Prof Md PhD, Principal Investigator — CH. Charles Perrens
Locations (1):
- Centre Hospitalier CHARLES PERRENS, Bordeaux, Gironde, France

REFERENCES:
- [Result] Petry NM, Blanco C, Auriacombe M, Borges G, Bucholz K, Crowley TJ, Grant BF, Hasin DS, O'Brien C. An overview of and rationale for changes proposed for pathological gambling in DSM-5. J Gambl Stud. 2014 Jun;30(2):493-502. doi: 10.1007/s10899-013-9370-0. PMID 23526033
- [Result] Hasin DS, O'Brien CP, Auriacombe M, Borges G, Bucholz K, Budney A, Compton WM, Crowley T, Ling W, Petry NM, Schuckit M, Grant BF. DSM-5 criteria for substance use disorders: recommendations and rationale. Am J Psychiatry. 2013 Aug;170(8):834-51. doi: 10.1176/appi.ajp.2013.12060782. PMID 23903334
- [Result] O'Brien C. Addiction and dependence in DSM-V. Addiction. 2011 May;106(5):866-7. doi: 10.1111/j.1360-0443.2010.03144.x. Epub 2010 Oct 6. PMID 21477226